CLINICAL TRIAL: NCT00423371
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of EUFLEXXA™ for Treatment of Osteoarthritis (OA) of the First Carpometacarpal (CMC) Joint
Brief Title: Double-Blind,Randomized,Placebo-Controlled Efficacy & Safety Study of EUFLEXXA™ for Treatment of OA of the First CMC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-02
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Osteoarthritis
Keywords: first Carpometacarpal (CMC) Joint
MeSH Terms: conditions — Osteoarthritis; Capillary Malformations, Congenital, 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUFLEXXA™ (Experimental)
  Interventions: Device: sodium hyaluronate
- Placebo (Placebo Comparator)
  Interventions: Device: placebo

INTERVENTIONS:
Device: sodium hyaluronate — EUFLEXXA™ is supplied in a single-dose syringe containing 20 mg/2 ml of 1% sodium hyaluronate. Each subject will receive three single dose injections into the target first CMC joint on study weeks 0, 2 and 4.
  Other Names: EUFLEXXA™
  Arms: EUFLEXXA™
Device: placebo — Placebo is supplied in a disposable prefilled glass syringe. Each single-dose syringe will contain 2 mL of phosphate buffered saline. Each subject will receive three single dose injections into the target first CMC joint on study weeks 0, 2 and 4.
  Arms: Placebo

SUMMARY:
This multicenter, double-blind, randomized, parallel-group, active-controlled trial will be performed in approximately 80 subjects with chronic idiopathic osteoarthritis (OA) of the first carpo-metacarpal joint (CMC).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥40 years of age
2. Pain due to primary OA of the first CMC joint present for at least half the days of the previous month AND a mean combined pain score ≥ 30 mm out of 100 mm of the 5 pain questions on the AUSCAN Index Pain Subscale (See Appendix 1)
3. A series of X-rays confirming OA of the first CMC joint of the target thumb obtained at screening with a stage of 2, 3, or 4 according to Grading Scale in Appendix 3.
4. Ability and willingness to use only acetaminophen as the analgesic (rescue) study medication

   * The acetaminophen dose must not exceed 4 grams/day (4000 mg)
   * If subject has known chronic liver disease, the maximum dose of acetaminophen must not exceed 2 grams/day (2000 mg)
   * The subject must be willing and able to discontinue acetaminophen at least 24 hours prior to all study-specific visits
   * The study specific acetaminophen provided will only be used for thumb/joint pain.
5. Willingness and ability to complete efficacy and safety questionnaires and ability to read and understand study instructions
6. Signed study-specific Subject Informed Consent Form

Exclusion Criteria:

1. Any major injury to the target thumb within the 6 months prior to the Screening Visit
2. Anyone having Carpal Tunnel Syndrome (CTS), DeQuervain's tenosynovitis, trigger finger, or a ganglion cyst of the target hand ONLY IF there is evidence of extreme atrophy AND two-point average discrimination is greater than 10-mm, OR if the pain from these conditions renders the subject unable to objectively assess OA pain in the target hand
3. Any surgery to the target joint within the 12 months prior to the Screening Visit
4. Regular use of assistive devices such as a cane or crutch or a CTS brace
5. Concomitant rheumatic disease (rheumatoid arthritis, lupus arthropathy, psoriatic arthritis)
6. History of chondrocalcinosis in the target joint
7. Gout exacerbation in any joint in the past 6 months
8. X-ray findings of acute fractures, severe loss of bone density, and/or severe bone or joint deformity in the target joint
9. Significant target joint infection or skin disorder/infection within the 3 months prior to study enrollment
10. Known hypersensitivity to acetaminophen, EUFLEXXA™, or Phosphate Buffered Saline solution
11. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period
12. Recurrent medical history of severe allergic or immune-mediated reactions or other immune disorders
13. Current treatment or treatment within the previous 2 years prior to the Screening Visit for any malignancy unless specific written permission is provided by the Sponsor (excluding basal cell or squamous cell carcinoma of the skin)
14. Active liver disease based on liver profile of AST, ALT, and conjugated bilirubin >2 times the upper limit of normal
15. Renal insufficiency based on serum creatinine >2.0 mg/dL
16. Any clinically significant laboratory value based on clinical history that the Investigator feels may affect the study evaluation
17. Any intercurrent chronic disease or condition that may interfere with the completion of the 6-month follow-up of the study, such as liver disease, severe coronary disease, drug abuse, disordered mental state, or other clinically significant condition
18. Current alcoholism, and/or any known current addiction to pain medications
19. Any clinically significant finding that would place the subject at health risk, impact the study, or affect the completion of the study
20. Any psychiatric illness that would prevent comprehension of the details and nature of the study
21. Participation in any experimental device study within 6 months prior to the Screening Visit, or an experimental drug study within 1 month prior to the Screening Visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean change in pain scores as reported by the patient on the AUSCAN Index pain subscale | weeks 0 and 26

SECONDARY OUTCOMES:
Mean change in stiffness and function scores as reported by the patient on the AUSCAN Index stillness and function subscale | weeks 0 and 26
Change in Patient Global Assessment of Symptoms measured by 100mm visual analog scale (VAS) | Weeks 0 and 26
Number of tablets of rescue medication used between visits | Weeks 0 and 26

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- All Florida Orthopedic Association, St. Petersburg, Florida, United States